CLINICAL TRIAL: NCT01635049
Title: Correlating Time-Lapse Parameters Detected by the Eeva™ System With Comprehensive Chromosome Screening Results,Implantation and Live Birth
Brief Title: Correlating Time-Lapse Parameters Detected by the Eeva™ System With Comprehensive Chromosome Screening Results
Acronym: CCS
Status: Completed | Type: Observational
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-AUX-004
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Infertility
Keywords: in vitro fertilization; assisted reproduction techniques; noninvasive imaging of embryos; time lapse imaging of embryos; traditional morphological grading of embryos; prediction of blastocysts; infertility; preimplantation genetic diagnosis; comprehensive chromosome screening
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women undergoing IVF treatment and CCS: •Women undergoing fresh IVF treatment and undergoing CCS, as recommended based on medical need by the clinical site reproductive endocrinologist.

SUMMARY:
The purpose of this research study protocol is to collect imaging data on embryos followed to blastocyst stage (Day 5-6) and correlate Eeva System parameters with comprehensive chromosome screening (CCS) results, implantation and live birth.

DETAILED DESCRIPTION:
The present study was designed to determine if there is a correlation between the Eeva System parameters and CCS results. Embryos will be selected for transfer based on CCS results and morphology. The Clinical site will have no access to the Eeva analysis at the time of the transfer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≤43 years of age.
* Women undergoing fresh IVF treatment using her own eggs or donor eggs and undergoing CCS, as recommended based on medical need by the clinical site reproductive endocrinologist.
* Fertilization using only ejaculated sperm (fresh or frozen) - no surgically retrieved sperm.
* Willing to have all 2PN embryos monitored by Eeva
* Not previously enrolled in this study.
* No concurrent participation in another clinical study.
* Willing to comply with study protocol and procedures and able to speak English.
* Willing to provide written informed consent.

Exclusion Criteria:

* BMI ≥ 40
* Prior IVF cycle with < 4 x 2PN
* Diminished ovarian reserve as demonstrated by any one of the following:

  * BAFC < 6 at time of cycle start
  * Maximum prior FSH > 15
  * AMH < 0.5

Max Age: 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women undergoing fresh IVF treatment and undergoing CCS, as recommended based on medical need by the clinical site reproductive endocrinologist.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Eeva time-lapse parameters and CCS | 5-6 days
  Analyse the correlation of time-lapse parameters collected by the Eeva System and comprehensive chromosome screening (CCS) results.

SECONDARY OUTCOMES:
Correlation of time-lapse parameters collected by the Eeva System and implantation rate. | 6 weeks
Correlation of time-lapse parameters collected by the Eeva System and clinical pregnancy rate | 6 weeks
Correlation of time-lapse parameters collected by the Eeva System and ongoing pregnancy rate | 7 - 8 weeks
Correlation of time-lapse parameters collected by the Eeva System and delivery rate | live birth
Correlation of time-lapse parameters collected by the Eeva System and spontaneous miscarriage rate | live birth
Correlation of time-lapse parameters collected by the Eeva System and multiple pregnancy rate | live birth

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, Jr., MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (2):
- United States (2):
  - Reproductive Medicine Associates of New Jersey, Morristown, New Jersey
  - Reproductive Medicine Associates of New York, New York, New York

REFERENCES:
- See also: Auxogyn, Inc. website — http://www.auxogyn.com